CLINICAL TRIAL: NCT05230251
Title: Radioligand fOr locAl raDiorecurrent proStaTe cancER
Acronym: ROADSTER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Glenn Bauman (Other)
Collaborators: London Health Sciences Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Glenn Bauman, Radiation Oncologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GB11498
Record Dates: First submitted 2022-01-19; First posted 2022-02-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Dose Radiation (HDR) arm (Active Comparator): Patients in the HDR arm will receive two fractions of HDR brachytherapy. HDR brachytherapy will be administered as per local practice and as previously described. All procedures will be conducted under general anesthesia in a dedicated brachytherapy suite using transrectal three dimensional ultrasound for image guidance. For all HDR fractions at least 10Gy will be delivered to the entire prostate with a boost to 13.5Gy to the involved prostate as determined by biopsy and PSMA PET/MRI results. In instances of multi-focal/diffuse involvement of the prostate, the entire prostate will receive 13.5Gy/fraction (respecting OAR constraints).
  Interventions: Radiation: High Dose Radiation
- Lutetium Arm (Experimental): Patients in Lutetium Arm will receive 1 cycle of 177Lu-PSMA radioligand therapy plus 1 fraction of HDR brachytherapy.
  Interventions: Drug: 177Lu-PNT2002; Radiation: High Dose Radiation

INTERVENTIONS:
Drug: 177Lu-PNT2002 — Men randomized to receive 177Lu-PSMA will receive 1 cycle of 177Lu-PSMA at a dose of 6.8MBq administered intravenously 2 weeks prior to the planned HDR administration in the Department of Nuclear Medicine as per local practice for the administration of therapeutic radiopharmaceuticals and consistent with good practices.
  Other Names: [Lu-177]-PNT2002 Injection
  Arms: Lutetium Arm
Radiation: High Dose Radiation — HDR brachytherapy will be administered as per local practice. All procedures will be conducted under general anesthesia in a dedicated brachytherapy suite using transrectal three dimensional ultrasound for image guidance. For all HDR fractions at least 10Gy will be delivered to the entire prostate with a boost to 13.5Gy to the involved prostate as determined by biopsy and PSMA PET/MRI results. In instances of multi-focal/diffuse involvement of the prostate, the entire prostate will receive 13.5Gy/fraction.

SUMMARY:
Approximately 50-60% of men undergoing salvage brachytherapy post cancer recurrence to the prostate have the disease controlled at 5 years. This study aims to integrate a local treatment to the prostate (brachytherapy) with a treatment involving 177Lutetium (Lu)- Prostate-Specific Membrane Antigen (PSMA) therapy. Differently than brachytherapy, 177-Lutetium-PSMA is thought to have its effect not only to the cancer cells within the prostate, but also to cancer cells located elsewhere in the body. Thus, the idea here is that by adding 177Lutetium (Lu)- PSMA early in the course of treatment we may be able to inactivate potential metastatic cells outside the prostate, while the prostate cancer within this organ still treated by the combination of brachytherapy and 177-Lutetium-PSMA.

DETAILED DESCRIPTION:
Surgery or radiation are common treatments for a prostate cancer that is confined to the prostate gland itself. After radiation treatment, a significant minority of patients (about one third) progress with cancer persistence or cancer regrowth (also known as local recurrence). Patients with local recurrent prostate cancer are eligible for additional treatments directed at the prostate. Prostate Specific Membrane Antigen (PSMA) is protein that is present in high quantities on prostate cancer and radioactive chemical "probes" against PSMA can identify those men with prostate cancer recurrence that is isolated to the prostate.

These radioactive probes can also be used to treat prostate cancer using high energy radioactive materials such as 177-Lutetium (Lu). A standard of care for the treatment of locally recurrent prostate cancer is the use of internal radiation (brachytherapy) delivered through needles inserted into the prostate from the outside. While brachytherapy allows high repeat doses of radiation to be given to the prostate and cancer, there is the potential to injury nearby structures such as the bladder and rectum. 177-Lu PSMA potentially provides a way to give an even more focused treatment to the cancer in the prostate (as well as treat any microscopic cancer that might be outside the prostate). In this study we will test the safety of integrating 177-Lu PSMA into the treatment of locally recurrent prostate cancer in combination with brachytherapy.

A total of 6 men per group (total=12) will be used in the first phase of this project to establish feasibility and safety of the combined treatment. Eligible participants will be chosen randomly to get one cycle of 177-Lu-PSMA treatment followed by brachytherapy treatment or the standard treatment of two brachytherapy treatments without 177-Lu-PSMA. All men will have biopsies (a small piece of tissue) and blood and urine samples taken at the time of the second brachytherapy treatment to compare markers of radiation effect from the first treatment with either 177-Lu-PSMA or brachytherapy. Toxicity assessment and Quality of Life questionnaires will be done at 6 weeks and 6 months after treatment to determine safety. Feasibility will be determined by the proportion of men in whom the treatment is delivered as planned. Provided safety and feasibility are established with the first 12 men, the study will continue to include 15 men per arm (30 men in total).

By developing a new treatment option for men with local recurrence after radiation, ROADSTER will be impactful for this group of men where existing treatments can carry significant side effects and are successful only about half the time.

ROADSTER trial is designed to involve two of the Lawson programs i.e. Imaging and Cancer and the trial participants will be treated in both departments. This inter-disciplinary collaboration is the key to answer the study question.

ELIGIBILITY:
Inclusion Criteria:

* Men with prostate adenocarcinoma treated with prior primary radiotherapy at least 2 years previously
* Biochemical failure according to the Phoenix criteria(Roach et al. 2006)
* PSMA PET demonstrating isolated uptake (SUV>3) within the prostate
* Biopsy confirmation of local recurrence within the prostate
* Not currently experiencing genitourinary (GU) or gastrointestinal (GI) Grade 3 or higher toxicity associated with prior treatment
* Adequate marrow function (Absolute neutrophil count ≥ 1.5 x 109/L -Platelet count ≥ 100 x 109/L

  -Hemoglobin ≥ 90 g/L with no transfusions in the past 2 weeks)
* Adequate renal function: Estimated creatinine clearance ≥ 30 ml/min according to Cockroft Gault equation:

  (140 - age) x (weight in kg) / 72 x (serum creatinine)
* Adequate liver function: Total bilirubin < 1.5 x upper limit of normal (ULN). Alanine aminotransferase (ALT) < 3.5 x ULN
* No contraindication to treatment with [177Lu-PSMA Agent]
* No contraindication to MRI
* No contraindication to therapy with high dose rate brachytherapy under general anaesthetic

Exclusion Criteria:

* Does not meet eligibility criteria
* Prior ablative radiotherapy to the prostate (prior HDR or LDR brachytherapy or SBRT/SABR to prostate)
* Documented extraprostatic or distant recurrence on PSMA PET
* Consent not obtained or declines randomization
* Declines HDR salvage or not fit for HDR salvage procedure
* Concurrent use of hormone therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As prostate cancer is a disease of male sex, the research project is inherently targeted to this population of patients.
Enrollment: 3 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy | At 24 weeks post treatment
  As a proof of concept study the primary endpoint will be feasibility and safety. Feasibility will be defined as the ability to complete all study interventions up to and including the 6 month assessment. Safety will be defined as no Grade >3 toxicity up to and including the 6 months assessment.

SECONDARY OUTCOMES:
Response rate to treatment | Preintervention and T=24 weeks
  Response rate to treatment will be measured by serial Prostate Specific Antigen (PSA) with response classified as a >50% decrease compared to pre-treatment PSA levels.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bauman, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendez LC, Dhar A, Laidley D, Moussa M, Gomez JA, Chin J, Lee TY, Thiessen JD, Hoover D, Surrey K, Helou J, Velker V, Correa RJ, D'Souza D, Bayani J, Bauman G. The use of Lutetium-177 PSMA radioligand therapy with high dose rate brachytherapy for locally recurrent prostate cancer after previous definitive radiation therapy: a randomized, single-institution, phase I/II study (ROADSTER). BMC Cancer. 2023 Apr 20;23(1):362. doi: 10.1186/s12885-023-10851-0. PMID 37081426